CLINICAL TRIAL: NCT02355314
Title: Doppler-based Renal Resistive Index in Assessing Renal Dysfunction Reversibility in ICU Patients
Acronym: R2D2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1208184; ANSM (Other: 2013-A00044-41)
Record Dates: First submitted 2015-01-22; First posted 2015-02-04 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Acute Kidney Injury
Keywords: ICU patients; Doppler-based renal
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ICU patients requiring mechanical ventilation (Experimental)
  Interventions: Other: Doppler-based renal; Biological: blood sample and urine sample

INTERVENTIONS:
Other: Doppler-based renal — Doppler-based renal : day 0 and day 3
Biological: blood sample and urine sample — blood sample and urine sample : day 0 and day 3

SUMMARY:
Acute kidney injury (AKI) is common in intensive care unit (ICU) patients and remains associated with a dismal prognosis. The diagnosis of AKI relies on functional criteria (oliguria and serum creatinine elevation), which carry several important limitations. Additionally, the investigators lack biomarker that may predict short term renal prognosis.

Doppler-based renal resistive index (RI) measurement is a rapid and noninvasive investigative tool that may hold promise for early AKI detection in ICU patients or in differentiating transient from persistent AKI in selected critically ill patients. Although several studies have suggested adequate performance in predicting short-term reversibility of AKI, most of these studies were performed in limited patient samples. Additionally, a recent study has identified discrepant results regarding its diagnostic performance.

The main objective of this large prospective multicentre study is to assess diagnostic performance of Doppler-based renal resistive index in diagnosing persistent AKI in critically ill patients requiring mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Sinus rhythm
* Use of conventional mechanical ventilation

Exclusion Criteria:

* Refusal: patient, family or trusted person to participate in the study
* Renal artery stenosis known
* Pregnant
* Severe Chronic Renal Failure (clearance < 30 ml.min-1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2013-12; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Doppler-based renal resistive index | Day 0
  Doppler-based renal resistive index in diagnosing persistent AKI in critically ill patients requiring mechanical ventilation

SECONDARY OUTCOMES:
Doppler-based renal resistive index | Day 3
Dosages NGAL plasmatique, NGAL urinaire, IGFBP-7, TIMP-2 | Day 0
Dosages NGAL plasmatique, NGAL urinaire, IGFBP-7, TIMP-2 | Day 3
usual urinary indices (Fractional excretion of urea, fractional excretion of sodium, ratio U / P urea ratio U / P creatinine) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Carine LABRUYERE, Chef de projet, Study Chair — URCIP
Locations (5):
- France (5):
  - CHU Avicenne, Bobigny
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHU Saint-Louis, Paris
  - Chu de Saint Etienne, Saint-Etienne
  - CHRU de Strasbourg, Strasbourg

REFERENCES:
- [Derived] Schnell D, Bourmaud A, Reynaud M, Rouleau S, Merdji H, Boivin A, Benyamina M, Vincent F, Lautrette A, Leroy C, Cohen Y, Legrand M, Morel J, Terreaux J, Darmon M. Performance of renal Doppler to predict the occurrence of acute kidney injury in patients without acute kidney injury at admission. J Crit Care. 2022 Jun;69:153983. doi: 10.1016/j.jcrc.2021.12.017. Epub 2022 Jan 21. PMID 35074631
- [Derived] Saade A, Bourmaud A, Schnell D, Darmon M; R2D2 Study Group. Performance of Doppler-Based Resistive Index and Semiquantitative Renal Perfusion in Predicting Persistent Acute Kidney Injury According to Operator Experience: Post Hoc Analysis of a Prospective Multicenter Study. Crit Care Med. 2022 Apr 1;50(4):e361-e369. doi: 10.1097/CCM.0000000000005372. PMID 34678845
- [Derived] Darmon M, Bourmaud A, Reynaud M, Rouleau S, Meziani F, Boivin A, Benyamina M, Vincent F, Lautrette A, Leroy C, Cohen Y, Legrand M, Morel J, Terreaux J, Schnell D. Performance of Doppler-based resistive index and semi-quantitative renal perfusion in predicting persistent AKI: results of a prospective multicenter study. Intensive Care Med. 2018 Nov;44(11):1904-1913. doi: 10.1007/s00134-018-5386-3. Epub 2018 Oct 5. PMID 30291377